CLINICAL TRIAL: NCT00769366
Title: Randomized, Controlled Study on Short-term Psychotherapy After Acute Myocardial Infarction: The Step-in-AMI Trial (Short TErm Psychotherapy IN Acute Myocardial Infarction)
Brief Title: Randomized, Controlled Study on Short-term Psychotherapy After Acute Myocardial Infarction
Acronym: STEP-IN-AMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Filippo Neri General Hospital (Other)
Responsible Party: Principal Investigator, Christian Pristipino, MD, Head of Research and Training section, Interventional Cardiology Unit, San Filippo Neri General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008
Record Dates: First submitted 2008-10-07; First posted 2008-10-09 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Acute Myocardial Infarction
MeSH Terms: interventions — Psychotherapy; Nutrition Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psychotherapy (Experimental): Psychotherapy and medical therapy
  Interventions: Behavioral: Psychotherapy
- Control (Active Comparator): Optimal medical therapy
  Interventions: Drug: Medical therapy

INTERVENTIONS:
Behavioral: Psychotherapy — humanistic-existential psychotherapy conducted in individual and group meetings
  Arms: Psychotherapy
Drug: Medical therapy — Optimal medical therapy after Acute myocardial infarction
  Arms: Control

SUMMARY:
Psychosocial factors play an important role in the pathophysiology of acute myocardial infarction (AMI), but it is not known if psychotherapy is beneficial after the contemporary treatment of AMI consisting of medical and interventional therapy.

The investigators have designed a randomized, controlled study to assess the effects of short-term psychotherapy (STP) on the clinical outcomes of patients who have undergone an emergency percutaneous coronary intervention (PCI) post-AMI.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to San Filippo Neri Hospital for AMI and treated with primary or urgent PCI.
* Primary PTCA is performed up to 12 hours after the beginning of chest pain in cases of STEMI, while patients with NSTEMI are enrolled if urgent PTCA is being performed within 48 hours of the onset of chest pain.
* Only patients in whom complete revascularization is achieved are being enrolled in the study.

Exclusion Criteria:

* Patients with psychiatric disorders or disability, cognitive impairment, or other life-threatening conditions are being excluded from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2005-06-02; Primary Completion 2011-11-01 (Actual); Study Completion 2016-11-01 (Actual)

PRIMARY OUTCOMES:
The cumulative incidence of new cardiological events and the occurrence of new medical pathologies | 5 years

SECONDARY OUTCOMES:
Incidence of re-hospitalisations | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- San filippo Neri Hospital, Rome, Italy

REFERENCES:
- [Derived] Pristipino C, Roncella A, Pasceri V, Speciale G. Short-TErm Psychotherapy IN Acute Myocardial Infarction (STEP-IN-AMI) Trial: Final Results. Am J Med. 2019 May;132(5):639-646.e5. doi: 10.1016/j.amjmed.2018.12.025. Epub 2019 Jan 17. PMID 30659815
- [Derived] Roncella A, Pristipino C, Cianfrocca C, Scorza S, Pasceri V, Pelliccia F, Denollet J, Pedersen SS, Speciale G. One-year results of the randomized, controlled, short-term psychotherapy in acute myocardial infarction (STEP-IN-AMI) trial. Int J Cardiol. 2013 Dec 10;170(2):132-9. doi: 10.1016/j.ijcard.2013.08.094. Epub 2013 Sep 8. PMID 24239154